CLINICAL TRIAL: NCT06507475
Title: Real World Effectiveness of Oral Semaglutide in Thailand Patients With Type 2 Diabetes: an Observational, Multicentre, Retrospective Cohort Study REAL-world Effectiveness of Oral Semaglutide In a Cohort of Thai patientS With Type 2 Diabetes treatED With Oral Antidiabetic Medications (REALISED) Study
Brief Title: Real World Effectiveness of Oral Semaglutide in Thailand Participants With Type 2 Diabetes
Acronym: REALISED
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9924-7830; U1111-1294-2999 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Semaglutide: Participants diagnosed with type 2 diabetes (T2D) who had initiated once-daily oral semaglutide during the target selection period of April 2022 to December 2023 and have not previously been treated with injectable glucose-lowering medication in routine clinical practice.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants treated with commercially available oral semaglutide according to local label and to routine clinical practice at the discretion of the treating physician.
  Other Names: Rybelsus

SUMMARY:
This study aims to describe the effectiveness of oral semaglutide on glycemic control and body weight control and describe characteristics of type 2 diabetes (T2D) adult patients who are being treated with oral semaglutide in Thailand. Data of eligible patients with T2D will be collected via electronic medical record or paper-format chart review to assess the effectiveness of oral semaglutide. Total study duration for the individual patient will be six months from baseline. The study duration expands within the window period will be 12 months from baseline which will be the optional visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult Thai male or female patients aged greater than or equal to (≥) 18 years.
* Diagnosed with T2D either through International Classification of Diseases (ICD) code or by physician's description such as documentation in the medical record, and who have not previously been treated with injectable glucose-lowering medication.
* At least one recent or closest Glycated Haemoglobin (HbA1c) test value available and documented less than or equal to 12 weeks prior to the initiation of oral semaglutide.
* Had initiated oral semaglutide for diabetes during the target selection period of April 2022 to December 2023. All required data for collection should already be accessible prior to the initiation of data collection.
* Treated with oral semaglutide for at least 6 months without interruption or discontinuation.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study (if applicable).
* Participants with any diagnosis of type 1 diabetes (T1D).
* Medical records documenting prior or ongoing treatment with injectable glucose-lowering treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with type 2 diabetes (T2D) who had initiated once-daily oral semaglutide during the target selection period of April 2022 to December 2023 and have not previously been treated with injectable glucose-lowering medication in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2024-09-07 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Glycated Haemoglobin (HbA1c) | Baseline (week 0), end of study (week 26)
  Measured in percentage-point of HbA1c.

SECONDARY OUTCOMES:
Absolute Change in Body Weight | At or within 12 months prior to baseline (week 0), end of study (week 26)
  Measured in kilograms.
Relative Change in Body Weight | At or within 12 months prior to baseline (week 0), end of study (week 26)
  Measured as percentage change in body weight.
Age of Participants | At baseline (week 0)
  Measured in years.
Percentage of Participants Assessed for Age | At baseline (week 0)
  Measured in percentage of participants.
Number of Participants Assessed for Gender (Male/Female) | At baseline (week 0)
  Measured in participants.
Percentage of Participants With Smoking History (Never, Previous, Current) | At baseline (week 0)
  Measured in percentage of participants.
Diabetes Duration of Participants | At baseline (week 0)
  Measured in years.
Percentage of Participants With Reasons to Initiate Oral Semaglutide Treatment | At baseline (week 0)
  Reasons will be categorized as: Improve glycemic control; Weight reduction; Address cardiovascular risk factors; Other. Measured in percentage of participants.
Body Weight | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  Measured in kilograms.
Diabetes Related Co-morbidities (modified Charlson Comorbidity Index [mCCI] Category) | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  The modified Charlson Comorbidity Index is a commonly used scale for assessing morbidity. It predicts the mortality for a patient who may have a range of comorbidities. It is based on comorbid conditions with varying assigned weights, resulting in a composite score. Each condition is assigned a score of 1, 2, 3, or 6, depending on the risk of dying associated with each one. Scores are summed to provide a total score to predict mortality. A score of zero indicates that no comorbidities were found, the higher the score, the higher the predicted mortality rate is.
  Measured in score on scale.
Fasting Plasma Glucose | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  Measured in milligrams per deciliter (mg/dL).
Post Prandial Glucose | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  Measured in milligrams per deciliter (mg/dL).
Diabetes Medications: Type of Drugs Class | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  Measured in participants.
Diabetes Medications: Number | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  Measured in number of diabetes medications.
Diabetes Medications: Dosage | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
Waist Circumference | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  Measured in centimeters.
Body Mass Index | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  Measured in kilograms per square meter (kg/m^2).
Blood Pressure (systolic/diastolic) | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  Measured in millimeters of mercury (mmHg).
Estimated Glomerular Filtration Rate (eGFR) | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  Measured in milliliters per minute (ml/min).
Creatinine | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  Measured in milligrams per deciliter (mg/dL).
Lipid profile: Low-density Lipoprotein Cholesterol (LDL), Non-high-density Lipoprotein Cholesterol (non-HDL), High-density Lipoprotein Cholesterol (HDL), Very Low Density Lipoprotein (VLDL), Total Cholesterol and Triglycerides | At or within 12 months prior to baseline (week 0) to optional visit (week 52-62)
  Measured in milligrams per deciliter (mg/dL).
Percentage of Participants Achieveing Glycated Haemoglobin (HbA1c) Less Than 7 Percentage (%) | At or within 12 months prior to baseline (week 0), end of study (week 26) and optional visit (week 52-62)
  Measured in percentage of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital_Nephrology, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com